CLINICAL TRIAL: NCT05144230
Title: Collection of Electronic Health Records (EHR) for Validation of Artificial Intelligence Based Tool for Data Quality Assessment
Brief Title: Healthy Data: Improving Health Information Quality Using Intelligent Systems
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Obinwa Ozonze, Principal Investigator, University of Portsmouth
Other Study IDs: UP717295
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Data Quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Electronic Health Record Systems (EHR) play an integral role in healthcare practice, enabling health organisations to collect, access and manage data more consistently. There is also a great deal of interest in using EHR data to improve decision-making and accelerate medical interventions. However, like all information systems, they are prone to data quality problems such as incomplete records, values outside normal ranges and implausible relationships. These problems are expected to become more prevalent as more organisations adopt electronic health record systems, aggregate, share and explore health data. The investigators believe current efforts to improve health data quality can be made more effective if backed by appropriate technology in the form of a readily accessible intelligent tool. Building on this, the investigators developed an Artificial Intelligence (AI) tool for automating data quality assessment of health data. In this study, the investigators evaluate the AI tool using a real-world dataset.

DETAILED DESCRIPTION:
The main aim of this study is to assess the reliability and utility of an AI tool in identifying data quality dimensions of interest for secondary use of health data, including completeness, conformance and plausibility. In assessing this tool, this study will retrospectively analyse data captured during routine clinical care and identify records containing listed data quality dimensions. This study will also assess the consistency of the AI tool in generating and executing data quality checks.

ELIGIBILITY:
Inclusion Criteria:

* No specific exclusion criteria

Exclusion Criteria:

* No specific exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient records captured by Portsmouth Hospitals University National Health Service Trust (PHU) between 01/01/2020 and 31/12/2020
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Data quality dimensions prevalence | 12 months, between 01/01/2020 and 31/12/2020
  The number of patient records identified by the AI tool with completeness, conformance and plausibility violations
Consistency of AI tool | 2 months, through study completion
  Consistency of AI tool in generating measures for detecting data quality dimensions
Validity of AI tool detection | 2 months, through study completion
  Validity of data quality dimensions identified by the AI tool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahn MG, Callahan TJ, Barnard J, Bauck AE, Brown J, Davidson BN, Estiri H, Goerg C, Holve E, Johnson SG, Liaw ST, Hamilton-Lopez M, Meeker D, Ong TC, Ryan P, Shang N, Weiskopf NG, Weng C, Zozus MN, Schilling L. A Harmonized Data Quality Assessment Terminology and Framework for the Secondary Use of Electronic Health Record Data. EGEMS (Wash DC). 2016 Sep 11;4(1):1244. doi: 10.13063/2327-9214.1244. eCollection 2016. PMID 27713905